CLINICAL TRIAL: NCT01657513
Title: Production of Antibodies Against Tnf-alfa Blockers in Patients With Psoriasis
Brief Title: TNF-alfa Inhibitors and Antibody Production in Patients With Psoriasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: The Michaelsen Foundation (Unknown); Pfizer (Industry)
Responsible Party: Principal Investigator, Peter Jensen, MD, University Hospital, Gentofte, Copenhagen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-2-2012-001; H-2-2012-001 (Registry Identifier: Ethics committee of the Capital Region of Denmark)
Record Dates: First submitted 2012-07-30; First posted 2012-08-06 (Estimated); Last update posted 2012-08-06 (Estimated); Status verified 2012-08

CONDITIONS: Psoriasis
Keywords: psoriasis; treatment failure; tnf-alfa
MeSH Terms: conditions — Psoriasis | interventions — Adalimumab; Etanercept; Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- tnf-alfa treatment (infliximab, adalimumab, or etanercept) (Experimental): This arm includes all the patients of the study. They are patients who are start treatment with a tnf-alfa blocking drug
  Interventions: Drug: subjects will receive either infliximab, adalimumab or etanercept

INTERVENTIONS:
Drug: subjects will receive either infliximab, adalimumab or etanercept — The subjects receive treatment with a tnf-alfa blocking according to the official guidelines for the particular drug.
  The study subjects will receive treatment with one drug only -
  1. infliximab or
  2. adalimumab or
  3. etanercept
  The consulting dermatologist decides which drug to use according to official guidelines
  Other Names: infliximab; adalimumab; etanercept

SUMMARY:
TNF alfa blockers are widely used for treatment of severe psoriasis. These biologics are well-tolerated with few side effects.

Unfortunately not all patients respond adequately to treatment with tnf alfa blockers. Some do not respond at all while others respond initially but gradually lose effect despite increased dose and more frequent administration.

The cause of treatment failure is largely unknown and it may be production of tnf-alfa neutralizing antibodies. This has been demonstrated in patients with rheumatoid arthritis and inflammatory bowel disease who lost response after treatment with tnf-alfa blockers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age above 18
* Psoriasis
* Indication for treatment with tnf alfa blocking drug
* Written informed consent obtained

Exclusion Criteria:

* Severe psychiatric disorder
* No indication for treatment with tnf-alfa blocking drug
* Pregnancy
* Breastfeeding
* No written informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
change in concentration of tnf-alfa antibodies in serum | 3, 6, and 12 months after start of tnf-alfa blocking agent
  Measurement (ELISA) of concentration of tnf-alfa neutralizing antibodies

SECONDARY OUTCOMES:
change in severity of psoriasis, PASI | 3, 6, and 12 months after start of tnf-alfa blocking agent
  severity of psoriasis assessed by PASI
Presence of psoriatic arthritis | 3, 6, and 12 months after start of tnf-alfa blocking agent
  Does the patient have psoriasis arthritis
change in dermatology life quality index (DLQI) | 3, 6, and 12 months after start of tnf-alfa blocking agent
  psoriasis severity assessed by the dermatology life quality index (DLQI)
height (cm) | 3 months
  subject´s height in centimeters
change in weight (kg) | 3, 6, and 12 months after start of tnf-alfa blocking agent
  subjects weight in kilograms

OTHER OUTCOMES:
assessment of change in concentrations of other biomarkers of interest in psoriasis | 3, 6, and 12 months after start of tnf-alfa blocking agent
  Collection of 3 ml of serum which are kept at -80 degrees celcius for later analysis of future biomarkers of interest

CONTACTS AND LOCATIONS:
Overall Officials: Lone Skov, MD, PhD, Study Director — Copenhagen University Hospital Gentofte, Department of Skin and Allergies; Mona Ståhle, MD, PhD, Principal Investigator — Karolinska Institute, Department of Medicine
Locations (2):
- Copenhagen University Hospital Gentofte, Department of Skin and Allergies, Hellerup, Denmark
- Karolinska Institute, Department of Medicine, Stockholm, Sweden